CLINICAL TRIAL: NCT07302672
Title: Humanistic Continuing Care Via WeChat for Patients Undergoing Thermal Ablation of Papillary Thyroid Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ming-an Yu (Other)
Responsible Party: Sponsor-Investigator, Ming-an Yu, Head of department of intervention medicine, China-Japan Friendship Hospital
Organization: China-Japan Friendship Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2509008
Record Dates: First submitted 2025-11-29; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Papillary Thyroid Carcinoma
Keywords: papillary thyroid carcinoma; thermal ablation; humanistic care; continuity care; Wechat; anxiety; quality of life
MeSH Terms: conditions — Thyroid Cancer, Papillary; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Personnel responsible for evaluating the primary or secondary outcome measures remain unaware of the participants' group assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Humanistic Continuing Care via WeChat (Experimental)
  Interventions: Behavioral: Humanistic Continuing Care via WeChat
- Usual Care (No Structured WeChat Program) (Active Comparator)
  Interventions: Procedure: Usual Care (No Structured WeChat Program)

INTERVENTIONS:
Behavioral: Humanistic Continuing Care via WeChat — Description: Structured, humanistic peri-operative nursing program delivered through WeChat in addition to routine care. Components: pre-procedure needs assessment and expectation setting; brief coping skills coaching (e.g., paced breathing); intra-procedure step-by-step explanations, reassurance, and comfort measures; post-procedure education, recovery guidance, and psychosocial support; symptom monitoring with red-flag escalation; medication/wound-care and appointment reminders; on-demand messaging during service hours; optional caregiver engagement.
  Delivery & Schedule: Nurse-led. One pre-procedure session; intra-procedure support on the day of ablation; post-procedure WeChat check-ins at least weekly plus on-demand messaging for 12 weeks. Fidelity tracked via standardized checklists.
  Arm(s): Experimental - Humanistic Continuing Care via WeChat.
  Arms: Humanistic Continuing Care via WeChat
Procedure: Usual Care (No Structured WeChat Program) — Participants receive standard peri-operative nursing and institutional discharge materials, including routine pre-procedure counseling, standard intra-procedure monitoring, printed/posted instructions for home care, and follow-up per usual practice (e.g., clinic visit or routine phone call). They may contact the clinic using standard channels as needed, but there is no scheduled, structured WeChat outreach or humanistic continuing-care protocol.
  Arms: Usual Care (No Structured WeChat Program)

SUMMARY:
The goal of this clinical trial is to test whether human-centered nursing care lowers emotional distress and improves quality of life for people who are awake during thyroid thermal ablation. The procedure uses local anesthesia, so participants remain awake and may feel tense. Human-centered care focuses on emotional support, clear communication, comfort, and follow-up, and it may improve the experience and recovery for patients.

The main questions are:

Does human-centered nursing care reduce emotional distress levels in patients undergoing thyroid thermal ablation?

Does human-centered nursing care improve patient quality of life after thyroid thermal ablation?

If there is a comparison group: Researchers will compare human-centered nursing care to usual nursing care to see if human-centered care leads to lower emotional distress and higher quality of life.

Participants will:

Receive either human-centered nursing care or usual nursing care.

Complete questionnaires before, during, and after the procedure to measure emotional distress, quality of life, pain, and satisfaction with care.

Have their vital signs and quality of life tracked during and after the procedure.

Have their adherence to care plans and any complications monitored.

The main outcomes are emotional distress levels and quality of life. Other outcomes include pain and vital signs during the procedure, satisfaction with care, and complication rates. Results may guide better care for people undergoing small, minimally invasive treatments while awake.

ELIGIBILITY:
Inclusion Criteria:

* Age 16-60 years; scheduled for thyroid thermal ablation
* Papillary thyroid carcinoma (PTC)
* Number of target lesions <= 3
* Largest lesion diameter <= 2 cm; clinical stage T1N0M0 by imaging
* Awake and able to cooperate under local anesthesia

Owns a smartphone and can use WeChat

Exclusion Criteria:

* Serious medical comorbidities or cognitive impairment that precludes participation
* Prior thyroid surgery or thermal ablation
* Unwilling or unable to join the WeChat group or complete postoperative follow-up

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in emotion distress from baseline to post-procedure (HADS) | From enrollment to the end of treatment at 3 months
Change in the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 scores from baseline to 3 months | From enrollment to the end of treatment at 3 months
Change in Thyroid Cancer-Specific Quality of Life Questionnaire scores from baseline to 3 months | From enrollment to 3 months after end of treatment

SECONDARY OUTCOMES:
Intraoperative pain intensity (Visual Analog Scale) | Intraoperative period (during the procedure)
  Pain intensity during the procedure will be assessed using a Visual Analog Scale (VAS; 0-100 mm, where 0 indicates no pain and 10 indicates the worst imaginable pain). A single VAS score will be recorded during the intraoperative period.
Patient satisfaction with nursing care (Newcastle Satisfaction with Nursing Scale, NSNS) | Postoperative Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided
Undecided at this time; a final decision about IPD sharing will be made after publication in consultation with the institution's data governance and ethics committees.